CLINICAL TRIAL: NCT06937671
Title: Randomized Trial of Cold EMR Compared to Hybrid Cold EMR.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Shah,Tilak, Medical Doctor, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-126
Record Dates: First submitted 2025-04-11; First posted 2025-04-22 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-04

CONDITIONS: Polyp of Colon; Endoscopic Mucosal Resection
Keywords: EMR; Cold EMR; Hybrid EMR; Endoscopic mucosal resection
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold EMR (Active Comparator): Control group patients that receive standard cold EMR treatment.
  Interventions: Procedure: Cold EMR
- Hybrid cold EMR (Experimental): Intervention group patients. Patients will receive hybrid EMR treatment.
  Interventions: Procedure: Hybrid EMR

INTERVENTIONS:
Procedure: Cold EMR — Cold EMR with cold forceps (regular or jumbo forceps) removal of any visible neoplasia that cannot be ensnared.
  Arms: Cold EMR
Procedure: Hybrid EMR — Cold EMR with hot avulsion of any visible residual neoplasia within the resection bed, in addition to precise APC of the fibrotic bands that may harbor invisible neoplasia within the resection bed.
  Arms: Hybrid cold EMR

SUMMARY:
The goal of this randomized clinical trial is to learn if a combination of hot and cold EMR technique is associated with a lower risk of polyp recurrence without increasing the risk of complication when removing large polyps.

Participants will undergo EMR and return for a follow-up endoscopy in 3-6 months to check for polyp recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age 18 years or older)
* Polyp size of at least 20 mm
* - Morphology: Flat or superficially raised polyp morphology (i.e., Paris classification 1s, 0-IIa or 0-IIb, or a combination of the above)

Exclusion Criteria:

* Polyps with previous failed resection attempts or polyp recurrence
* Suspected deep submucosal invasion on endoscopic assessment of surface mucosal pit pattern (Kudo V or NICE 3 pattern) or histologically confirmed malignancy (invasive adenocarcinoma)
* Polyps with nodules too large (>1-1.5cm) for the use of a cold snare
* Inflammatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence of polyps | 3-6 months after the procedure
  Recurrence of polyps confirmed by biopsy at the site of EMR on follow-up colonoscopy

SECONDARY OUTCOMES:
Adverse events | 3-6 months after the procedure
  Composite of clinically important adverse events: (1) Perforation requiring hospitalization or surgery (2) Bleeding associated with at least 2-gram Hb drop or hospitalization or Intervention (3) Post-polypectomy syndrome requiring hospital admission
Polyp recurrence rates | 3-6 months after EMR procedure
  Recurrence of polyps confirmed by biopsy at the site of EMR on follow-up colonoscopy
Cost benefit analysis | 3-6 months after the procedure
  - Cost-benefit analysis includes the costs of additional hospitalizations related to post-procedure complications and the cost of additional colonoscopies required to follow up treatment of recurrence. Costs will be calculated from a Medicare perspective.
Subgroup polyp recurrence rate | 3-6 months after the procedure
  - Recurrence rates in the subgroup of patients with visible residual neoplasia after snare resection before utilizing forceps or cautery resection/ablation

CONTACTS AND LOCATIONS:
Overall Officials: Tilak Shah, M.D., Principal Investigator — Cleveland Clinic Florida (Weston Hospital)
Locations (2):
- United States (2):
  - Cleveland Clinic Weston, Weston, Florida
  - Cleveland Clinic, Cleveland, Ohio